CLINICAL TRIAL: NCT05961995
Title: Acute and Long-term Effects of App-delivered Heartfulness Meditation on Psychological Outcomes and the Endocannabinoid Signaling System in Cyclic Vomiting Syndrome
Brief Title: Heartfulness Meditation (HFM) in Cyclic Vomiting Syndrome (CVS)
Acronym: HFM-CVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Thangam Venkatesan, Principal Investigator, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022H0078
Record Dates: First submitted 2023-04-05; First posted 2023-07-27 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cyclic Vomiting Syndrome
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFN Meditation (Experimental): Subjects will complete guided meditation sessions 3 x a week for six weeks delivered in the app via video, as well as pre- and post-meditation psychological state assessments.
  Interventions: Behavioral: Heartfulness meditation

INTERVENTIONS:
Behavioral: Heartfulness meditation — Heartfulness meditation is a secular, specific, guided meditation technique that includes progressive relaxation with a concentrated focus on the heart. The HFN meditation will last 30 minutes. There will be a prescribed progressive relaxation technique which will last for ~ 5-10 minutes followed by the heart-based meditation.

SUMMARY:
Cyclic vomiting syndrome (CVS) is a chronic disorder of gut-brain interaction (DGBI) characterized by episodes of vomiting often triggered by stress. CVS affects 2% of the population and has a disproportionate negative impact on patients and the healthcare system. Although gastrointestinal symptoms are prominent, most patients have comorbid anxiety, depression, high degrees of psychological distress, and other negative cognitive traits that adversely affect health-related quality of life (HRQoL). This is independent of typical measures of severity of CVS and warrants treatment. Recent guidelines recommend a biopsychosocial model of care incorporating techniques like meditation to mitigate stress and improve psychological outcomes in CVS. One potential approach to improve these outcomes is the use of heartfulness (HFN) meditation.

Heartfulness meditation is a secular, specific, guided meditation technique that includes progressive relaxation with a concentrated focus on the heart. It is offered virtually and is free-of charge ensuring no barriers to broad application in clinical practice. A pilot study incorporating HFN meditation in CVS significantly reduced psychological distress, perceived stress, and improved coping strategies, sleep quality, and HRQoL. Other data also show that HFN meditation improves overall well-being and reduces perceived stress. However, there are significant gaps in our understanding of the mechanism underlying HFN meditation and its effects on patient outcomes.

The endocannabinoid signaling system (ECSS) is activated by stress exposure and functions through multiple neuroendocrine responses to mitigate the negative effects of stress. We examined the role of the ECSS in CVS and found that endocannabinoids were not elevated during an acute CVS episode. This lack of a response in the ECSS during an acute CVS episode, which is characterized by panic, intense nausea and vomiting is striking, given that the ECSS is typically activated by stress exposure. This may reflect an underlying dysfunction of the ECSS in CVS and impaired stress responsivity. Given these data and our preliminary findings of the beneficial effects of HFN meditation, our central hypothesis is that HFN meditation will increase circulating endocannabinoids in CVS and that this will be correlated with a reduction in anxiety and other psychological outcomes and overall quality of life.

We propose to test our hypothesis with the following specific aims

Specific Aim 1a: Conduct a prospective study to elucidate the acute effects of HFN meditation on the ECSS in CVS. We will measure circulating endocannabinoids and related lipids immediately before and after HFN meditation.

1b: Correlate indices of ECSS with state anxiety and mood pre-and post-HFN meditation. We will measure state anxiety and mood with validated tools including the State Trait Anxiety Inventory (STAI) and Profile of Mood States (POMS) which evaluates tension, depression, anger, vigor, fatigue, and confusion.

Hypothesis: HFN meditation will acutely increase circulating endocannabinoids which will be correlated with a reduction in state anxiety and improvement in mood.

Specific Aim 2: Determine the long-term effects of a 6-week HFN meditation program on ECSS and correlate with psychological outcomes including psychological distress, STAI scores, sleep quality, and HRQoL. We will measure these outcomes with validated tools including the Brief Symptom Inventory (BSI), STAI, Pittsburgh Sleep Quality Index (PSQI), and PROMIS quality of life questionnaires.

Hypothesis: A regular HFN meditation practice over 6 weeks will further augment ECSS, and this will be correlated with an improvement in psychological outcomes such as psychological distress, sleep, mood and HRQoL.

DETAILED DESCRIPTION:
Research Design

Design: We will conduct a single-arm uncontrolled pilot study with 40 patients. Patients aged 18-80 years diagnosed with CVS based on Rome criteria will be eligible to participate.

Exclusion criteria: 1. Major psychiatric illness such as schizophrenia, bipolar disease, and major depression or anxiety that is not controlled with medication or requiring inpatient care within the past year 2. History of suicidal attempt/ideation in the past year 3. Cognitive impairment that precludes the ability to meditate 4. Inability to sit for at least 30 minutes 5. Severe cardiopulmonary diseases, malignancy, or renal failure on dialysis 6. Other organic gastrointestinal diseases or systemic diseases including but not limited to inflammatory bowel disease and chronic liver diseases 7. Pregnancy at the time of enrollment 8. BMI < 18 or >35 9. Regular cannabis use (defined as daily or near-daily cannabis use) and 10. Individuals with significant prior meditation experience (continuous meditation practice for ≥ 3 months within a year prior to the study).

Patients will come for 2 study visits. Subjects will complete guided meditation sessions 3 x a week for six weeks delivered in the app via video, as well as pre- and post-meditation psychological state assessments. The app will automatically document meditation compliance, and study staff will be able to remind patients if compliance is inadequate. The app will be HIPAA compliant and only study staff will have access to PHI.

Study procedures:

Screening of potential study participants via web form and telephone. Study visit 1: Enrollment and baseline visit: Consenting, web app orientation, completion of baseline questionnaires, completion of first 30 min. meditation session using the app, with pre- and post-meditation blood draw.

Intervention: Six weeks of self-administered heart-focused meditation, consisting of 3 meditation sessions per week, each approximately 30 minutes in length, delivered via video guidance in the app.

Study visit 2: End-of-study visit. Completion of end-of-study questionnaires via the web app, final 30-min meditation session during the visit with pre-post session blood draw.

The web-based app: This will be custom-designed research (Heartsapp), which can be used on any smartphone or electronic tablet. The existing Heartsapp created by the HFN Institute will be modified and will be compliant with HIPAA privacy rules. Dr. Olafur Palsson at the University of North Carolina at Chapel Hill will serve as a consultant who has pioneered such applications. The HFN Institute has committed to modifying their existing app for research.

Psychological outcomes These will be measured using validated tools including the a. State-Trait-Anxiety Inventory (STAI)31 and profile of Mood States (POMS) c. Basic Symptom Inventory (BSI)33 at baseline, 3 and 6 weeks. Other parameters such as HRQOL (PROMIS), sleep quality (Pittsburgh Sleep Quality Index)35 and other measures of coping (COPE) will also be measured at these time points. Perceived intervention effectiveness will be assessed with a visual analog scale (VAS) ("0" not effective at all; "10" most effective imaginable) after intervention sessions at baseline and at end of study at 6 weeks.

Individual meditation protocol Subjects will be instructed to be seated in a comfortable position in a neutral room. They are instructed not to lie down during the session as this may promote sleep. The HFN meditation will last 30 minutes. There will be a prescribed progressive relaxation technique which will last for ~ 5-10 minutes followed by the heart-based meditation. This period of relaxation prepares them for the focused meditation. During the focused meditation, subjects will be instructed to bring their focus to the heart. They will be asked to make a gentle supposition that there is a source of light in the heart. They will be given specific instructions on how to deal with their thoughts. Unlike other forms of meditation, HFN meditation does not focus on the breath. Subjects are simply instructed to breathe normally during the session. The remainder of the meditation session (20 minutes) will be in silence. After the meditation session, the instructor will indicate that the session is ending. Participants will be asked to gently open their eyes, observe their inner state, and write down their observations.

Statistical analysis We expect that circulating endocannabinoids will increase immediately following HFN meditation and that this will be correlated with a reduction in state anxiety and improvement in mood. We will use a paired t-test to compare the circulating endocannabinoids at baseline (20 minutes prior) and 5-10 minutes post-intervention and compare patients' baseline and post-intervention psychological outcomes (STAI score for anxiety and POMS score for mood states) All of the baseline outcomes will also be compared with their values after the 6-week meditation checking further effects of the intervention. Transformation of the outcomes may be needed if the normality assumption is violated.

Blood collection procedures A small intravenous catheter will be placed in the forearm or wrist area and blood samples will be obtained (20 minutes prior) and 5-10 minutes post-intervention in the seated position. During each collection,10ml of blood will be collected in one red top serum-separating tube and will be refrigerated immediately. Plasma will be separated from blood by centrifugation and stored at -80 °C until analysis.

Endocannabinoid concentrations and related lipids Deuterated 2-AG and AEA will be added to the sera, followed by lipid extraction using solid phase columns as previously detailed.25 Concentrations of AEA, 2-AG, PEA, and OEA will be quantified by isotope dilution following measurement using atmospheric pressure, chemical ionization liquid chromatography/mass spectrometry (LC-APCI-MS) as described previously.14

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 80 years of age
* Diagnosed with CVS based on Rome criteria

Exclusion Criteria:

* Major psychiatric illness such as schizophrenia, bipolar disease, and major depression or anxiety that is not controlled with medication or requiring inpatient care within the past year
* History of suicidal attempt/ideation in the past year
* Cognitive impairment that precludes the ability to meditate
* Inability to sit for at least 30 minutes
* Severe cardiopulmonary diseases, malignancy, or renal failure on dialysis
* Other organic gastrointestinal diseases or systemic diseases including but not limited to inflammatory bowel disease and chronic liver diseases
* Pregnancy at the time of enrollment
* BMI < 18 or >35
* Regular cannabis use (defined as daily or near-daily cannabis use) and
* Individuals with significant prior meditation experience (continuous meditation practice for ≥ 3 months within a year prior to the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venkatesan T, Hillard CJ, Ayer L, Arumugam S, Culp S, Vyas M, Gofar K, Petrova A, Palsson OS. Acute and Long-Term Effects of App-Delivered Heartfulness Meditation on Psychological Outcomes and the Endocannabinoid Signaling System in Cyclic Vomiting Syndrome. Clin Transl Gastroenterol. 2024 Jul 1;15(7):e00711. doi: 10.14309/ctg.0000000000000711. PMID 38713142

RESULTS

PARTICIPANT FLOW:
Groups:
- HFN Meditation: Subjects will complete guided meditation sessions 3 x a week for six weeks delivered in the app via video, as well as pre- and post-meditation psychological state assessments.
  Heartfulness meditation: Heartfulness meditation is a secular, specific, guided meditation technique that includes progressive relaxation with a concentrated focus on the heart.
Period: Overall Study
Arm/Group | HFN Meditation
Started | 45
Completed | 30
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- HFN Meditation: Patients aged 18-80 years diagnosed with cyclic vomiting syndrome based on Rome criteria who meet the eligibility criteria were assigned for the 6 week heartfulness meditation sessions.
Arm/Group | HFN Meditation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 23
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: State-Trait-Anxiety Inventory (STAI) (18) and Profile of Mood States (POMS)
Description: The primary outcomes were state and trait anxiety and mood states, measured using the State-Trait-Anxiety Inventory (STAI) and Profile of Mood States (POMS) respectively. The STAI-S evaluates current feelings of apprehension, tension, nervousness, and worry. The scale consists of two 20-item subscales and four rating categories including very much so, moderately so, somewhat and not at all. Scores for STAI range from 20 to 80. Higher scores indicate great anxiety, lower scores indicate no or low anxiety.
  The POMS is a 35-item validated questionnaire that assesses mood states of tension, depression, anger, vigor, fatigue and confusion. There is a variation in the range of scores for each subscale, with the lowest being 0 and the highest 60. A lower score indicates a better mood, and vice versa. Total score is calculated by summing the totals for the negative subscales and then subtracting the totals for the positive subscales with a higher score indicating worse mood disturbance.
Time Frame: 6 weeks
Population: Patients aged 18-80 years diagnosed with CVS who meet the Rome criteria
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HFN Meditation
Number analyzed (Participants) | 30
score on a scale
  Baseline (week 1) State anxiety | 34.59 (10.48)
  Week 3 State anxiety | 35.05 (10.19)
  week 6 State anxiety | 26.27 (6.95)
  baseline (Week 1) Trait Anxiety | 41.67 (15.02)
  Week 3 Trait Anxiety | 39.76 (11.98)
  week 6 Trait Anxiety | 36.10 (11.73)
  Baseline (week 1) POMS | 54.46 (14.44)
  Week 3 POMS | 48.75 (9.28)
  Week 6 POMS | 46.43 (9.67)

2. Secondary Outcome: Brief Symptom Inventory (BSI) - General Severity Index (GSI), Health-related Quality of Life (PROMIS), Sleep Quality (Pittsburgh Sleep Quality Index) Coping (COPE), and Visual Analog Scale (VAS) Effectiveness Score
Description: BSI-GSI scores are converted to area t-scores, with a mean of 50 and a standard deviation of 10. A higher t-score indicates greater psychological distress, whereas a lower t-score indicates less psychological distress. PROMIS scores in the clinical sample are reported as T-scores, with a mean of 50 and a standard deviation of 10. Higher T-scores for PROMIS Mental and PROMIS Physical indicate better mental and physical health respectively. PSQI sleep quality scores have a total minimum and maximum score of 0 and 21. A score of 0-5 is considered a good quality of sleep, whereas 6- 21 is considered a poor quality of sleep. COPE for religion and spirituality minimum score of 2 indicates no or limited use of spirituality or religion as a coping tool, whereas a maximum score of 8 indicates greater reliance on spirituality or religion as a coping strategy. VAS ranges from 0 to 10, a higher and lower VAS score indicates an increased and decreased perceived effectiveness respectively.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HFN Meditation
Number analyzed (Participants) | 30
score on a scale
  BSI GSI BASELINE | 57.86 (10.59)
  BSI GSI WEEK 3 | 55.68 (9.68)
  BSI GSI WEEK 6 | 54.21 (9.56)
  PROMIS Baseline-Mental | 46.63 (9.44)
  PROMIS week 3-Mental | 46.89 (7.81)
  PROMIS week 6-Mental | 49.87 (8.33)
  PROMIS Baseline-Physical | 46.61 (9.37)
  PROMIS week 3-Physical | 48.2 (9.81)
  PROMIS week 6-Physical | 49.76 (8.29)
  Sleep quality (PSQI)-Baseline | 1.21 (0.73)
  Sleep quality (PSQI)-Week 3 | 0.96 (0.88)
  Sleep quality (PSQI)-Week 6 | 0.71 (0.76)
  COPE- Religion/spirituality -Baseline | 3.76 (2.02)
  COPE- Religion/spirituality-Week 3 | 5.07 (1.77)
  COPE - Religion/spirituality- Week 6 | 5.31 (1.56)
  VAS effectiveness score - baseline | 6.40 (1.50)
  VAS effectiveness score - Week 6 | 6.40 (1.83)

ADVERSE EVENTS:
Time Frame: Adverse event were collected at Baseline (week 1) and Week 6
Description: Participants were thoroughly briefed on potential risks and provided with contact information for study coordinators who can offer support and guidance. During each in-person visit and follow up phone calls, adverse events are reviewed and documented in the participant's binder. The study team including the principal investigator assess/grade the findings and take the necessary steps to resolve them. A serious adverse event is promptly reported to the local IRB as per protocol.
Groups:
- Single Arm Study: We conducted a 6-week single-arm pilot study to assess the effects of Heartfulness meditation (HFM) in CVS using a custom-designed meditation app. Primary outcomes included state and trait anxiety and mood state changes pre- vs. post-meditation, and secondary outcomes were psychological distress, coping, sleep quality and Health-Related Quality of Life at baseline and weeks 3 and 6. Serum concentration of endocannabinoids N-arachidonylethanolamine (AEA) and 2-arachidonoylglycerol (2-AG) and related lipids were measured pre-and-post HFM at baseline and week 6.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
This was a single-arm study and the expectation of a positive response might have influenced the results and hence our findings need to be confirmed with randomized controlled trials. This intervention is not accessible to those without a smartphone but this represents <10% of the US population. We did not assess effects on CVS symptom frequency or healthcare utilization related to CVS as this was a 6-week trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT05961995/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT05961995/ICF_001.pdf